CLINICAL TRIAL: NCT00711958
Title: Double-blind, Randomized, Multicenter, Clinical Phase III Study to Evaluate the Efficacy and Safety of HX575 for the Treatment of Chemotherapy Associated Anemia in Cancer Patients
Brief Title: Study to Assess the Efficacy and Safety of HX575 in the Treatment of Chemotherapy Associated Anemia in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-31-INJ-11
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Anemia
Keywords: Chemotherapy associated anemia in cancer patients
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HX575 epoetin alfa Hexal AG (Experimental): HX575 (erythropoietin alfa of the Sponsor Hexal AG). Eligible patients to be randomized in ratio 2:1 and to be subcutaneously treated (solution for injection (s.c.)) for 12 weeks with HX575 in pre-filled syringes. The maximum weekly dose of HX575 was 300 IU/kg body weight to maintain hemoglobin levels in the therapeutic range. Application of the drug required at least once per week and allowed maximum three times per week.
  Interventions: Drug: HX575, solution for injection (s.c.)
- ERYPO® Janssen-Cilag (Active Comparator): ERYPO® Janssen-Cilag, Germany. Eligible patients were treated subcutaneously (solution for injection (s.c.)) with ERYPO® (Janssen-Cilag, Germany) in pre-filled syringes for 12 weeks.The maximum weekly dose of HX575 was 300 IU/kg body weight to maintain hemoglobin levels in the therapeutic range. Application of the drug required at least once per week and allowed maximum three times per week.
  Interventions: Drug: ERYPO®, Janssen-Cilag, solution for injection (s.c.)

INTERVENTIONS:
Drug: HX575, solution for injection (s.c.) — 1000, 2000, 4000, 8000 and 10.000 IU of rh erythropoiethin
  Other Names: Binocrit, Erythropoeitin alfa Hexal, Abseamed
  Arms: HX575 epoetin alfa Hexal AG
Drug: ERYPO®, Janssen-Cilag, solution for injection (s.c.) — 1000, 2000, 4000, 8000 and 10.000 IU of epoetin alfa
  Other Names: Eprex
  Arms: ERYPO® Janssen-Cilag

SUMMARY:
This is a randomized, double-blind, multicenter clinical phase III study involving about 105 cancer patients aged >18 years who are receiving palliative chemotherapy and who are suffering from chemotherapy associated anemia. A standard treatment group (ERYPO®) will be included to provide a reference reflecting current standard medical practice.

DETAILED DESCRIPTION:
Eligible patients were randomized to one of two different treatment groups (EPO HEXAL or ERYPO) in a 2:1 ratio. Patients received double-blind treatment for a period of 12 weeks. Following randomization the patients were treated subcutaneously with a dose of 150 IU/kg body weight of study drug three times per week. Dose adjustments to 300 IU/kg body weight three times per week were to be done if hemoglobin (Hb) increased <1.0 g/dL or the reticulocyte count increased <40,000 /μl after 4 weeks or if Hb increased <2.0 g/dL after 8 weeks of treatment. The primary endpoint was the Hb response in the EPO HEXAL group during weeks 5-12 of the study defined as absolute increase in Hb value of 2.0 g/dL from the mean value of the screening/baseline period in the absence of red blood cell transfusion during the preceding 4 weeks. For that purpose, Hb levels were measured at the weekly study visits by a central laboratory. Further parameters of treatment efficacy, safety and tolerability were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of solid tumors
* Patients who receive cyclic palliative chemotherapy with a cycle duration of 1 -4 weeks (for at least 12 weeks) during the study
* Patients with chemotherapy associated anemia (hemoglobin < 10.0 g/dl at screening)
* Life expectancy of at least 6 months Age: > 18
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2
* Serum ferritin greater or equal to 100 µg/l and/or saturated transferrin levels greater or equal to 20 %
* Adequate renal function (serum creatinine below or equal to 2.0 mg/dl)
* Adequate hepatic function (bilirubin < 1.5 times upper limit of normal range
* Patients with ability to follow study instructions, likely to complete all required visits and able to perform the quality of life assessment
* Written informed consent of the patient

Exclusion Criteria:

* Patients who receive curative intended chemotherapy
* Known primary or metastatic malignancy of the central nervous system
* Known primary or metastatic malignancy of bone marrow
* Primary hematologic disorder (e.g. myelodysplastic syndrome, sickle cell anemia, hematological malignancy, acute leukemia)
* Thrombotic events during the last 6 months
* Suspicion or known PRCA (pure red cell aplasia)
* Transfusion of white blood cells or packed red blood cells (more than 2 packs) within 4 weeks and any transfusion of white blood cells or packed red blood cells within 2 weeks prior to randomization (visit 0)
* Anemia due to overt bleeding or hemolysis within 2 weeks before screening
* Erythropoietin or Darbepoietin therapy within 8 weeks before screening, including any investigational form of erythropoietin (e.g. gene-activated erythropoietin, novel erythropoiesis stimulating protein)
* Radiation therapy during the study, radiation therapy induced anemia
* Therapy with cyclosporine
* Chemotherapy which causes predictable treatment with peripheral-blood progenitor therapy, e.g. G-CSF
* Clinical evidence of current uncontrolled hyperparathyroidism (serum parathyroid hormone >1500 pg/mL)
* Major surgery within 14 days prior to randomization
* Treatment with antiepileptics within the last 5 years
* Previously diagnosed HIV or acute hepatitis infection
* Uncontrolled hypertension, defined as a diastolic blood pressure measurement >110mm Hg during the screening period
* History of congestive heart failure (NYHA class III, IV)
* Unstable angina pectoris, active cardiac disease, cardiac infarction during the last six months before screening
* Evidence of acute infectious disease or serious active inflammatory disease within four weeks before screening (Visit -1) or during the screening/baseline period
* Known allergy to one of the ingredients of the test or reference products or hypersensitivity to mammalian-derived products
* Pregnancy, breastfeeding women or women not using adequate birth control measures
* Patients who participate simultaneously in another clinical study or who have participated in a study in the month preceding the start of this study or previously randomized to this study (except studies with approved medications in an approved indication, with an approved dosing regimen including approved treatment combinations)
* Suspicion of any non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-11; Primary Completion 2005-07 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vetter, Dr., Study Chair — Hexal AG
Locations (19):
- Germany (15):
  - Gemeinschaftspraxis Drs. Brudler, Heinrich, Bangerter, Augsburg
  - Gemeinschaftspraxis mit Schwerpunkt Hämatologie und Internistische Onkologie, Bad Soden
  - Poliklinik am Paritätischen Krankenhaus, Berlin
  - Schwerpunktpraxis für Brustkrankheiten und Gynäkologische Onkologie, Berlin
  - Oskar-Helene-Heim, Berlin
  - Praxis Drs. Marschner, Zeiss, Kirste, Freiburg im Breisgau
  - DRK-Krankenhaus, Luckenwalde
  - Praxis für Onkologie, Munich
  - Praxis Drs. Kowolik/Prechtl, Munich
  - Klinikum Nürnberg, 5. Medizinische Klinik Haus 12, Zimmer Nr. 13, Nuremberg
  - Gemeinschaftspraxis, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Tübingen Medizinische Klinik 1, Tübingen
  - Gemeinschaftspraxis für internistische Onkologie, Velbert
  - Praxis für internistische Onkologie, Weiden
- Romania (4):
  - Oncologic Institute, Cluj-Napoca
  - Country hospital Oradea, Oradea
  - County Hospital Satu-Mare, Satu Mare
  - Oncomed SRL Timisoara, Timișoara

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 cancer centers, in Germany and Romania .
Pre-assignment Details: 2:1 randomization All 114 patients found eligible were randomized and treated (60 in Germany and 54 in Romania)
Period: Overall Study
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO® Janssen-Cilag
Started | 74 | 40
Completed | 41 | 17
Not Completed | 33 | 23
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Lack of Efficacy | 3 | 1
Not completed — Clinical deterioration | 1 | 0
Not completed — Adverse Event | 9 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 10 | 5
Not completed — Progression of disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: 50 patients found to have a major protocol violation , excluded from the ITT population only (31 and 19 in EPO HEXAL and ERYPO groups), none from the Safety Analysis population. Major deviations: early patient withdrawal (consent or due to AE), and lack of endpoint value in observation period (no Hemoglobin value over weeks 5 to 12)
Groups:
- Total: Total of all reporting groups
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO® Janssen-Cilag | Total
Number analyzed (Participants) | 74 | 40 | 114
Age, Customized [Count of Participants; unit: Participants]
  18-39 years | 3 | 3 | 6
  40-64 years | 43 | 18 | 61
  ≥65 years | 28 | 19 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 17 | 58
  Male | 33 | 23 | 56
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 36 | 18 | 54
  Germany | 38 | 22 | 60
most frequent site of primary malignancy [Count of Participants; unit: Participants]
  ovary | 17 | 7 | 24
  lung | 13 | 6 | 19
  pancreas | 5 | 4 | 9
  stomach | 4 | 4 | 8
  breast | 8 | 3 | 11
  other | 27 | 16 | 43

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of HX575 in the Treatment of Chemotherapy Associated Anemia
Description: Proportion of patients with a change in hemoglobin levels more than 2 g/dL under treatment with HX575, estimated between weeks 5-12.
Time Frame: 5-12 weeks
Population: Intention-to-treat population: patients with post baseline Hemoglobin value available
Measure: Count of Participants; unit: Participants
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO® Janssen-Cilag
Number analyzed (Participants) | 60 | 34
Participants | 37 | 15

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Treatment emergent adverse events were collected, starting from the day of study medication administration
Arm/Group | HX575 Epoetin Alfa Hexal AG | ERYPO® Janssen-Cilag
All-Cause Mortality (participants affected / at risk) | 18/74 | 12/40
Serious Adverse Events (participants affected / at risk) | 34/74 | 18/40
Other Adverse Events (participants affected / at risk) | 62/74 | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 Epoetin Alfa Hexal AG (N=74) | ERYPO® Janssen-Cilag (N=40)
Neoplasms malignant site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 6 (6)
Metastases to specified sites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Neoplasms unspecified malignancy and site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oncologic complications and emergencies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal neoplasms malignant NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stenosis and obstruction NEC (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 1 (1) | 2 (2)
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal and rectal ulcers and perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (excl infective) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal and small intestinal stenosis and obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcers and perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (excl infective) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernias (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhages (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (excl infective) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenic conditions (General disorders) | 4 (4) | 0 (0)
Febrile disorders (General disorders) | 0 (0) | 2 (2)
Implant and catheter site reactions (General disorders) | 2 (2) | 0 (0)
General signs and symptoms NEC (General disorders) | 1 (1) | 0 (0)
Pain and discomfort NEC (General disorders) | 1 (1) | 0 (0)
Renal failure and impairment (Renal and urinary disorders) | 2 (2) | 5 (5)
Urinary abnormalities (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal obstructive disorders (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal lithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular arrhythmias and cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Heart failures NEC (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic coronary artery disorders (Cardiac disorders) | 0 (0) | 2 (2)
Rate and rhythm disorders NEC (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular arrhythmias (Cardiac disorders) | 0 (0) | 1 (1)
Anaemias NEC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemias due to chronic disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Marrow depression and hypoplastic anaemias (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenias (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenias (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cholestasis and jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic failure and associated disorders (Hepatobiliary disorders) | 2 (2) | 0 (0)
Obstructive bile duct disorders (excl neoplasms) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diabetes mellitus (incl subtypes) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
General nutritional disorders NEC (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Potassium imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Total fluid volume decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower limb fractures and dislocations (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphoedemas (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism and thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular hypertensive disorders NEC (Vascular disorders) | 1 (1) | 0 (0)
Sepsis, bacteraemia and viraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infections (Infections and infestations) | 1 (1) | 0 (0)
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coma states (Nervous system disorders) | 1 (1) | 0 (0)
Disturbances in consciousness NEC (Nervous system disorders) | 1 (1) | 0 (0)
Retinopathies NEC (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 Epoetin Alfa Hexal AG (N=74) | ERYPO® Janssen-Cilag (N=40)
Nausea (Gastrointestinal disorders) | 17 (23) | 14 (25)
Vomiting (Gastrointestinal disorders) | 13 (16) | 9 (15)
Constipation (Gastrointestinal disorders) | 9 (13) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (3)
Asthenia (General disorders) | 15 (21) | 6 (7)
Pyrexia (General disorders) | 9 (15) | 4 (5)
Fatigue (General disorders) | 5 (5) | 6 (6)
Oedema peripheral (General disorders) | 5 (5) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 12 (16) | 7 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
leukopenia (Blood and lymphatic system disorders) | 4 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (5) | 3 (3)
iron deficiency (Metabolism and nutrition disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results stemming from the present trial can only be published if both the Coordinating investigator and the sponsor give their consent. Publications of subcollectives or center specific data are only possible if the whole study results have already been published.